CLINICAL TRIAL: NCT07196709
Title: Effect of High-power Laser Acupuncture on Fatigue and Proprioception in Chronic Non-specific Low Back Pain: A Randomized Controlled Trail
Brief Title: Effect of High-power Laser Acupuncture on Fatigue and Proprioception in Low Back Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Doaa Ayoub Elimy Mohammed, Lecturer of physical therapy for basic science department., faculty of physical Therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/005223
Record Dates: First submitted 2025-09-20; First posted 2025-09-29 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Chronic Nonspecific Low-back Pain
Keywords: low back pain; high-power laser acupuncture; fatigue; proprioception; Pain self-efficacy
MeSH Terms: conditions — Low Back Pain; Fatigue

STUDY DESIGN:
Intervention Model Description: high-power laser acupuncture and exercise therapy program
Who Masked: Participant, Outcomes Assessor
Masking Description: random generator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high-power laser acupuncture and the exercise program (Experimental): The patients will receive high-power laser acupuncture and the exercise program three times a week for 4 weeks.
  Interventions: Device: high-power laser acupuncture and the exercise program
- sham laser acupuncture and exercises program (Sham Comparator): The patients will receive sham acupuncture laser and the exercise program three times a week for four weeks.
  Interventions: Device: sham laser acupuncture and the exercises program

INTERVENTIONS:
Device: high-power laser acupuncture and the exercise program — The experimental group will receive high-power lasers, and the treatment will be performed at 15 acupuncture points: unilateral GV3, GV4, and GV5, and bilateral BL 20, BL23, BL24, BL25, BL40, and GB30. Exercises program: The patients will perform this exercise program in the form of: strengthening exercises for abdominal and back muscles; lumbar stabilization exercises; and stretching exercises
  Other Names: high-intensity laser acupuncture
  Arms: high-power laser acupuncture and the exercise program
Device: sham laser acupuncture and the exercises program — The patients will receive a sham laser acupuncture and the exercise program in the form of: strengthening exercises for abdominal and back muscles; lumbar stabilization exercises and stretching exercises.
  Other Names: sham laser acupuncture
  Arms: sham laser acupuncture and exercises program

SUMMARY:
To investigate the effect of high-intensity laser acupuncture on fatigue, proprioception, back pain and Pain self-efficacy in patients with chronic nonspecific low back pain (CNLBP).

DETAILED DESCRIPTION:
Chronic non-specific low back pain (CNSLBP) is a persistent back pain that affects people of all ages and significantly impacts individuals' functional activities. Fatigue and impaired proprioception are common complaints associated with CNSLBP, contributing to diminished physical performance and exacerbation of symptoms. While various treatment modalities exist, there is ongoing interest in exploring novel approaches to manage this condition effectively.Laser photobiomodulation (PBM) therapy is a noninvasive that stimulates cells, pain receptors, and the immune system and can cause analgesic effects. Recently, high-power lasers have been used for managing musculoskeletal dysfunction that allows for more energy deposition in deep tissues, resulting in both biological and thermal effects. High-power laser acupuncture (HPLA) has emerged as a promising intervention that combines the therapeutic effects of high-power laser therapy and the principles of acupuncture point stimulation on the body (acupoints) to induce physiological effect. However, there is limited evidence supporting this combined approach. For that, this study aims to investigate the effect of HPLA on fatigue, proprioception back pain and Pain self-efficacy in patients with CNSLBP. With this current randomized controlled trial, we seek to provide evidence-based insights into the potential effects of this combined approach on measurements of fatigue, proprioception, back pain and Pain self-efficacy.

ELIGIBILITY:
Inclusion Criteria:

* 1. The patients had CNSLBP with age from 20 to 40 years from both genders.

  2. Patients diagnosis with chronic low back pain without underlying pathological causes.

  3. The patients with chronic nonspecific low back pain more than 3months. Minimum pain intensity of 30 mm on the visual analogue scale (VAS) for pain, which ranges from 0 to 100 mm.

  4. Patients with BMI ranges between 18.5:29.9 kg/m2.

  5. The study populations must be willing to participate in the study

Exclusion Criteria:

1. Neurological, infectious diseases and systemic illness such as rheumatologic diseases,systemic lupus erythematosus, diabetes mellitus type I or II.
2. Psychiatric/mental deficit.
3. Patients who had a previous surgical history (within 6 months) will also excluded
4. participation in other treatment within the previous 3 month.
5. Pregnancy.
6. History of spinal fracture, tumor, osteoporosis

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
fatigue | up to six weeks
  Isokinetic dynamometer will be used for measuring fatigue of back muscles.
fatigue | up to six weeks
  The Biering-Sørensen test will be used for measuring fatigue of back muscles
proprioception | up to six weeks
  Isokinetic dynamometer will be used for assessing lumber proprioception

SECONDARY OUTCOMES:
Pain Intensity | up to six weeks
  The Visual Analogue Scale (VAS) will be used by the patient to mark his/her level of pain on a 0 to 100 millimeter line. Zero usually represents 'no pain at all,' whereas the upper limit represents 'the worst pain ever possible.' Higher scores represent worse pain intensity, and lower scores represent less pain.
Pain-Related Self-Efficacy | up to six weeks
  The Arabic version of the Pain Self-Efficacy Questionnaire (PSEQ-A) will be used to assess patients ' confidence in managing pain and performing daily activities. Higher scores reflect greater self-efficacy, indicating stronger confidence in coping with pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Doaa Ayoub Elimy, Giza, Egypt